CLINICAL TRIAL: NCT05164068
Title: Effect of an Informative Video Upon Anxiety and Stress in Patients Requiring an Oral Biopsy
Brief Title: Effect of an Informative Anxiety and Stress in Patients Requiring an Oral Biopsy
Acronym: Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Investigador principal Head Oral Medicine, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: adcobiusac 023-2021
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Anxiety ; Dental
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information video (Experimental): The experimental group likewise consisted of 60 individuals that received information about the biopsy procedure in video format
  Interventions: Behavioral: Information video
- Information face-to -face (No Intervention): The control group consisted of 60 patients that received face-to-face verbal information in a homogeneous and reproducible manner

INTERVENTIONS:
Behavioral: Information video — The video contents were clear and adapted to the characteristics of the population of Guatemala. The video provided a simple description of the biopsy, its risks and benefits, complications and general recommendations, and was presented preoperatively
  Arms: Information video

SUMMARY:
In clinical practice, patients scheduled for biopsy often suffer substantial stress before, during or after the procedure. In particular, most patients feel uncomfortable both with the procedure itself and with the idea of the results of the biopsy.

Providing adequate information is crucial, though there is no agreement as to which is the best way to present such information. Although verbal information provided by the professional is the most common scenario, the use of written information in the form of explanatory leaflets, as well as audio recordings or videos, has also been proposed The present study was carried out at the Dental School of Universidad de San Carlos (Guatemala) to evaluate the hypothesis that an audiovisual intervention providing information on oral biopsy is able to reduce patient anxiety and stress.

DETAILED DESCRIPTION:
A prospective, randomized clinical trial was carried out involving. A total of 120 patients were therefore finally randomized, following the Consort Statement guidelines, with the definition of two groups: a control group (n = 60) that received standard verbal information, and an experimental group (n = 60) that received information in the form of a video

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were a patient age of over 18 years and the presence of an oral lesion/s requiring biopsy.

Exclusion Criteria:

* Patients with decompensated systemic disorders, poor general condition, a history of psychiatric disease or psychoactive drug use were excluded, as were pregnant women and individuals failing to sign the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Anxiety level comparison biopsy with two preoperative information types | Baseline
  Modified Dental Anxiety Scale (MDAS) was used to assess anxiety levels. The Modified Dental Anxiety Scale (MDAS) consisted of 5 questions ranging from 5 (no anxiety) to 25 (highest anxiety level). Every patient was asked to mark his or her perceived dental anxiety level on the line.
Anxiety level comparison biopsy with two preoperative information types | 1 day of Final measure of the biopsy intervention
  Modified Dental Anxiety Scale (MDAS) was used to assess anxiety levels. The Modified Dental Anxiety Scale (MDAS) consisted of 5 questions ranging from 5 (no anxiety) to 25 (highest anxiety level). Every patient was asked to mark his or her perceived dental anxiety level on the line.

SECONDARY OUTCOMES:
Evaluate patient-reported pain levels | Baseline
  The Visual Analog Scale (VAS) will be used on a 0 to 10 scale, 0 being no pain at all and 10 being the worst pain imaginable.
Evaluate patient-reported pain levels | 1 day of final measure of the biopsy intervention
  The Visual Analog Scale (VAS) will be used on a 0 to 10 scale, 0 being no pain at all and 10 being the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CS, Wu SY, Yi CA. Association between Anxiety and Pain in Dental Treatment: A Systematic Review and Meta-analysis. J Dent Res. 2017 Feb;96(2):153-162. doi: 10.1177/0022034516678168. Epub 2016 Nov 16. PMID 28106507
- [Background] Caltabiano ML, Croker F, Page L, Sklavos A, Spiteri J, Hanrahan L, Choi R. Dental anxiety in patients attending a student dental clinic. BMC Oral Health. 2018 Mar 20;18(1):48. doi: 10.1186/s12903-018-0507-5. PMID 29558935